CLINICAL TRIAL: NCT07032467
Title: Examining the Relationship Between Social Media Addiction and Compulsive Exercise Behaviors in University Students
Brief Title: Social Media Addiction and Compulsive Exercise Behaviors
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: SMA-Exercise-1
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Social Media Addiction: Participants scoring 41-73 (No Addiction) or 74-106 (Mild Addiction) on the Social Media Addiction Scale (SMAS)
  Interventions: Other: Psychosocial and Behavioral Assessment
- High Social Media Addiction: Participants scoring 140-205 (High to Very High Addiction)
  Interventions: Other: Psychosocial and Behavioral Assessment

INTERVENTIONS:
Other: Psychosocial and Behavioral Assessment — Participants completed validated self-report questionnaires to assess levels of social media addiction and compulsive exercise behaviors. No therapeutic or experimental intervention was administered. Data were collected through surveys for observational analysis.

SUMMARY:
This cross-sectional study investigates the association between social media addiction levels and compulsive exercise behaviors among university students aged 18-24. Using validated self-report instruments, the study explores how increasing digital media engagement relates to exercise patterns and dependency traits, offering insights into the psychological-behavioral dynamics of young adults in the digital age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Between 18-24 years of age
* Spending at least 4 hours a day on social media
* Voluntarily participating in the study

Exclusion Criteria:

* Participants must be under 18 and over 24 years of age,
* Surf social media for less than 4 hours a day,
* Have a diagnosed psychiatric disorder

Ages: 18 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: University students aged 18-24 years residing in Istanbul, spending ≥4 hours daily on social media, with no psychiatric diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Social Media Addiction Score (SMAS) | Single assessment at baseline
  Social Media Addiction Scale (41 items, 4 subscales: preoccupation, mood modification, relapse, conflict)
  Scale Range: 41-205
  Scoring Categories:
  41-73: No Addiction
  74-106: Mild Addiction
  107-139: Moderate Addiction
  140-172: High Addiction
  173-205: Very High Addiction

SECONDARY OUTCOMES:
Compulsive Exercise Score (EXES) | Single assessment at baseline
  Tool: Exercise Addiction Scale (17 items, 3 factors: obsessive focus, social conflict, tolerance/passion)
  Scale Range: 17-85
  Scoring Categories:
  1-17: Normal
  18-34: Low Risk
  35-51: At Risk
  52-69: Addicted
  70-85: Highly Addicted

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided